CLINICAL TRIAL: NCT04366128
Title: Camrelizumab, Pegaspargase and Apatinib With Radiation Therapy for Stage IE/IIE Natural Killer /T-cell Lymphoma
Brief Title: Camrelizumab, Pegaspargase and Apatinib With Radiation Therapy for Stage IE/IIE ENKTL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rong Tao (Other)
Responsible Party: Sponsor-Investigator, Rong Tao, Associate director of department of hematology, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Organization: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XHLSG-NK-1902
Record Dates: First submitted 2020-04-25; First posted 2020-04-28 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Natural Killer/T-Cell Lymphoma, Nasal and Nasal-Type
Keywords: camrelizumab; apatinib; pegaspargase; radiotherapy; natural killer/T-cell lymphoma
MeSH Terms: interventions — Radiotherapy

STUDY DESIGN:
Intervention Model Description: Camrelizumab, apatinib and pegaspargase
Masking Description: Camrelizumab, apatinib and pegaspargase indution immunotherapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAPA indution immunotherapy (Experimental): CAPA regimen, repeat every 3 week for 4 cycles.
  Interventions: Drug: CAPA indution immunotherapy

INTERVENTIONS:
Drug: CAPA indution immunotherapy — 1. Camelirumab 200mg Intravenous injection on day 1.
  2. Apatinib 250mg taken orally once daily.
  3. Pegaspargase 2000U/m2 Intramuscular injection on day 1.
  Other Names: Radiotherapy

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of camrelizumab, apatinib, pegaspargase (CAPA) and as an intruction immunotherapy with radiotherapy as first-line treatment in patients with de novo stage IE/IIE extranodal natural killer/T-cell lymphoma, nasal type.

DETAILED DESCRIPTION:
Extranodal natural killer/T-cell lymphoma (ENKTCL), nasal type, is a rare subtype of non-Hodgkin lymphoma (NHL) with relatively high incidence in China. Radiotherapy alone for stage IE/IIE diseases has good response rate but with high relapse rates, ranging from 20-50%. The combination of chemotherapy and radiotherapy improved the long-term survival for patients with stage IE/IIE diseases. But the optimal treatment schedule has not been established. This study is designed with four cycles CAPA induction immunotherapy, followed by 50-56Gy radiotherapy as an approach for stage IE/IIE ENKTCL. The efficacy and safety of this treatment will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet the WHO 2016 diagnostic criteria for NK/T-cell lymphoma by biopsy histopathology, immunohistochemistry and EBER.
* The primary site is in the nasal cavity or upper gastrointestinal tract. The de novo diagnosed patient has at least one objective and evaluable lesion.
* Stage IE / IIE disease according to Lugano 2014 lymphoma staging system.
* ECOG score 0-3.
* The laboratory examination within 1 week before entering the group meets the following conditions:

  1. Blood routine test: neutrophil count≥1.0 × 10^9/L, Hemoglobin≥80g/L, Platelet≥50 × 10^9/L.
  2. Coagulation routine: plasma fibrinogen ≥ 1.0g / L.
  3. Liver function: Alanine aminotransferase, aspartate aminotransferase and total bilirubin ≤ 2 times the upper limit of normal value.
  4. Renal function: Creatinine is normal.
  5. Refers to oxygen saturation> 93%.
  6. Cardiac function: Left ventricular ejection fraction ≥50%, electrocardiogram does not suggest any acute myocardial infarction, arrhythmia or atrioventricular block above 1 degree
* Signed informed consent.
* Voluntarily follow the research protocol, follow-up plan, laboratory and auxiliary examinations.

Exclusion Criteria:

* accompanied with HCV or HIV infection, HBV-infected patients who also receive antiviral treatment are not excluded.
* Severe infection requires ICU treatment.
* Serious complications such as hemophagocytic syndrome, DIC, etc.
* Impairment of important organ functions: such as respiratory failure, chronic congestive heart failure with NYHA grade ≥3, decompensated liver or kidney dysfunction, hypertension and diabetes that cannot be controlled despite active treatment.
* Have a history of autoimmune diseases, have disease activity in the last 6 months, and are still taking oral immunosuppressive therapy within the past three months, with a daily dose of oral prednisone greater than 10 mg.
* Pregnant and lactating women.
* Those who are known to be allergic to drugs in the CAPA regimen.
* Patients with other tumors who need surgery or chemotherapy within 6 months.
* Other experimental drugs are being used.
* The investigators believe that other clinical conditions (including medical history or the presence of comorbidities) of the patient will significantly increase the risk of the subject when using the study treatment drugs.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-04-25 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Rate of complete response at week 24 | 24 weeks
  Rate of patients with complete response (CR) at week 24 evaluate by Lugano 2014 criteria

SECONDARY OUTCOMES:
Rate of overall response rate at week 24 | 24 weeks
  Rate of patients with complete response and partial response (ORR) at week 24 evaluate by Lugano 2014 criteria
Rate of overall survival at 2 years | 2 years
  overall survival rate (OS) of patients at 2 years
Rate of progression free survival at 2 years | 2 years
  progression free survival rate (PFS) of patients at 2 years
percent of adverse events | 2 years
  adverse events graded by NCI CTCAE Ver4.03

CONTACTS AND LOCATIONS:
Overall Officials: Rong Tao, MD, Principal Investigator — Xinhua Hospital, Shanghai Jiaotong University School of Medicine
Locations (3):
- China (3):
  - Sun Yat-sen University, Guangzhou, Guangdong
  - Shanghai Eye Ear Nose and Throat Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Department of Hematology, Xinhua hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No